CLINICAL TRIAL: NCT02262897
Title: Single Arm Phase II Clinical Trial to Investigate the Efficacy and Safety of Nab-paclitaxel as a Single Agent in the Small Cell Lung Cancer Patients With Extensive Disease and Failed to First Line/ Second Line Chemotherapy
Brief Title: The Efficacy and Safety of Nab-paclitaxel in Pretreated Patients With Extensive Disease of Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Shanghai Pulmonary Hospital, Tongji University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FK1401
Record Dates: First submitted 2014-09-23; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; chemotherapy; Nab-paclitaxel
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nab-paclitaxel single agent (Experimental): Nab-paclitaxel single agent, either in 130mg/m2 weekly regimen, d1,8,15 every 4 weeks or in 230mg/m2 d1 every 3 weeks
  Interventions: Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Nab-paclitaxel — Nab-paclitaxel weekly chemotherapy 130mg/m2, d1,8,15,every 4 week or Nab-paclitaxel chemotherapy once a time with a dose of 230 mg/m2 every 3 weeks
  Other Names: Albumin-bound paclitaxel， Abraxane

SUMMARY:
Patients with extensive disease(ED) small cell lung cancer is still have a dismal prognosis, even though the first line chemotherapy showing about 70% response rate. Most of the patients will relapse with in 6 months after the chemotherapy and the following therapy such as second line chemotherapy have a very limited efficacy to these patients. Currently, there is no standard 3rd line therapy for the patients with ED small cell lung cancer(SCLC).

As the investigators know, Nab-paclitaxel had showing promising efficacy in several cases report in the patients with SCLC, the aim of this clinical trial is to investigate the efficacy and safety of nab-paclitaxel as a single agent in the SCLC patients with extensive disease and failed to first line/ second line chemotherapy.

DETAILED DESCRIPTION:
Primary end point: Objective Response Rate(ORR)

Secondary end point:

Progression Free Survival(PFS), Overall Survival(OS), Side effects according to Common Terminology Criteria for Adverse Events(CTCAE) version 4.0 Quality Of Life(QOL) etc.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain of informed consent.
2. Male or female aged 18 years and over.
3. Histologically or cytologically confirmed small cell lung carcinoma.
4. Extensive disease before receive nab-paclitaxel.
5. Failed to previous chemotherapy, but the previous paclitaxel chemotherapy is not allowed.
6. World Health Organization (WHO) performance status (PS) of 0 to 2.
7. Females of child-bearing potential must have negative serum pregnancy test. Sexually active males and females (of childbearing potential) willing to practice contraception during the study.
8. Heart index values is in the range, as defined below, within two weeks of randomization:

   * Absolute neutrophils count(ANC)≥2.0×109/L
   * Platelets≥100×109/L
   * Serum bilirubin≤2×ULN; Aspartate transaminase(AST) and alanine transaminase (ALT) ≤2.5×ULN(≤5×ULN if liver metastases)
   * Creatinine clearance≥60ml/min
9. Measurable disease according to Response Evaluation Criteria in Solid Tumors(RECIST) criteria with at least one measurable lesion not previously irradiated.
10. Life expectancy ≥12 weeks.

Exclusion Criteria:

1. As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease).
2. Newly diagnosed Central Nervous System (CNS) metastases that have not yet been definitively treated with surgery and/or radiation.
3. Known severe hypersensitivity to nab-paclitaxel or any of the excipients of these products.Known severe hypersensitivity to pre-medications required for treatment with nab-paclitaxel doublet chemotherapy.
4. Prior treatment with paclitaxel.
5. Pregnant or lactating woman.
6. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ.
7. Life expectancy of less than 12 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | tumor assessment every 6-8 weeks after the initiation of chemotherapy, up to 24 months
  To evaluate Objective response rate every 6-8 weeks after the initiation of chemotherapy and before the completion of chemotherapy

SECONDARY OUTCOMES:
Progression free survival | 24 months
  PFS is evaluated in the 24 months since the treatment began
overall survival | 24 months
  evaluated in the 24th month since the treatment began
Side effects | 24 months
  evaluated in the 24th month since the treatment began according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Quality Of Life | 24 months
  evaluated in the 24th month since the treatment began

CONTACTS AND LOCATIONS:
Overall Officials: Guanghui Gao, Study Chair — Tongji University Affiliated Shanghai Pulmonary Hospital; Chunxia Su, Study Chair — Tongji University Affiliated Shanghai Pulmonary Hospital; Xiaoxia Chen, Study Chair — Tongji University Affiliated Shanghai Pulmonary Hospital; Wei Li, Study Chair — Tongji University Affiliated Shanghai Pulmonary Hospital
Locations (1):
- Shengxiang Ren, Shanghai, China